CLINICAL TRIAL: NCT05320445
Title: A Psychosocial Transitional Group to Improve Adaptation, Coping and Mental Health Outcomes Following Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4859
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-12

CONDITIONS: Musculoskeletal Injury; Traumatic Injury
Keywords: Group Therapy; Neuromusculoskeletal Traumatic Injury; Feasibility
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician analyzing the data will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supportive-expressive group therapy (Experimental): The SEGT is a six-module program where each session is approximately one hour, and is held twice a week over a three-week period. It is framed within social cognitive theory, whereby resilience to adversity (NMSK trauma in this instance) relies on personal enablement. Enablement serves to equip the individual with the personal resources to cultivate their self-efficacy and mastery and to select and construct environments that promote successful adaption.
  Interventions: Behavioral: Supportive Expressive Group Therapy
- Treatment as usual (No Intervention): The treatment as usual group will receive standard care only (which may include an individual psychiatric consultation).

INTERVENTIONS:
Behavioral: Supportive Expressive Group Therapy — The SEGT is a six-module program where each session is approximately one hour, and is held twice a week over a three-week period. It is framed within social cognitive theory, whereby resilience to adversity (NMSK trauma in this instance) relies on personal enablement. Enablement serves to equip the individual with the personal resources to cultivate their self-efficacy and mastery and to select and construct environments that promote successful adaption.
  Arms: Supportive-expressive group therapy

SUMMARY:
Traumatic physical injuries result in significant disability and a high proportion of survivors suffer from chronic pain and mental health disorders. A key predictor of good outcomes following trauma is "coping self-efficacy" - a person's belief that they can cope with life's challenges. Interventions that enhance coping self-efficacy post-injury are most likely to optimize recovery. However, these interventions are not standard approaches in rehabilitation settings.Our inter-disciplinary team will undertake a trial to assess the efficacy of supportive-expressive group therapy in rehabilitation inpatients who have had traumatic injuries. We wish to test whether persons who undergo the group therapy have significant improvements in coping self-efficacy compared to those receiving standard care. Sixty patients with traumatic injuries admitted to St. John's Rehab will be randomized to either supportive-expressive group therapy (n=30) or to standard rehabilitation (n=30). Additionally, up to 12 staff participants will be recruited.The goal of this project is to establish a gold standard for inpatient rehabilitation in the trauma NMSK injured population by widening the access to emotional wellbeing supports, which could translate into better physical, mental and social health in the community.

DETAILED DESCRIPTION:
Traumatic neuromusculoskeletal (NMSK) injuries result in significant disability and a high proportion of survivors suffer from chronic pain and mental health disorders. Inpatient acute care and rehabilitation are important treatments for patients after NMSK injury, however much of the work to ensure successful community participation occurs after discharge. A key mechanism for predicting outcomes following trauma is coping self-efficacy, therefore interventions that enhance coping self-efficacy post-NMSK injury are most likely to optimize recovery. However, these interventions are not standard approaches in rehabilitation settings.

Our inter-disciplinary team will undertake a feasibility randomized control trial (RCT) to assess the efficacy of supportive-expressive group therapy (SEGT) in NMSK injury rehabilitation inpatients. It is hypothesized that persons who undergo the SEGT will yield significant improvements in coping self-efficacy compared to those receiving standard care.

A prospective feasibility RCT design will be used to evaluate SEGT for NMSK injury rehabilitation inpatients compared to the standard rehabilitation for trauma patients at St John's Rehab (SJR). Sixty patients with an NMSK injury admitted to SJR will be randomized to either SEGT (n=30) or to standard rehabilitation (n=30). Additionally, up to 12 staff participants will be recruited to complete qualitative interviews/focus groups.

A repeated measures ANOVA will be used to detect differences on the outcome measures, which will include a group, time, and groups by time interaction term. Linear regression will be used to adjust for potential covariates of interest. A thematic content analysis will be used to analyze the qualitative data.

The long-term outcomes of this project is to establish a gold standard for inpatient rehabilitation in the trauma NMSK injured population by widening the access to emotional wellbeing supports, which could translate into better physical, mental and social health in the community.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking adults aged 18 years and older.
2. Admitted to SJR for inpatient rehabilitation.
3. Trauma-related peripheral nerve injury, muscle injury, amputation, and/or fracture(s).
4. Are medically stable.
5. Have no clinical suspicion of cognitive impairment or unstable severe mental health diagnosis (e.g. moderate/severe brain injury, schizophrenia, dementia, etc.).

Exclusion Criteria:

1. Are actively suicidal.
2. Are unable participate effectively in a group setting (e.g. actively using substances, exhibiting threatening behaviors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Participant recruitment | Through study completion, an average of 1 year.
  Number of participants who are recruited into the study and are contacted for assessments at set time intervals.
Questionnaire completion rates | Through study completion, an average of 1 year.
  Number of completed assessments
Treatment adherence | Through study completion, an average of 1 year.
  Number of participants who complete all 6 SEGT sessions
Number of participants contacted for follow up interview | At 1 month-post discharge for SEGT group]
  Number of participants contacted for follow up interview
Participant retention | At three months post-discharge for SEGT and control group
  Number of participants who complete the 3 month post-discharge assessments
Participant Retention | At one month post-discharge for SEGT group]
  Number of participants who complete 1 month post-discharge interview
Barriers and Facilitators to Group Participation | At one month post-discharge for SEGT group
  As discussed in qualitative interviews

SECONDARY OUTCOMES:
Change in Health-related quality of life | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  Short Form-36 Survey (SF-36): The SF-36 is the most widely used generic health-related QoL tool. The tool measures 8 domains including physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, social functioning, general mental health, role limitations due to emotional problems, and vitality. The minimum score is 0, and the maximum is 100. Higher scores on the measure are indicative of less disability.
Change in coping self-efficacy | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  Coping Self-Efficacy Scale (CSES): The CSES is a measures perceived self-efficacy for coping with challenges and threats. It is a 26-item measure rated using an 11-point scale with the anchors 0 (cannot do at), 5 (moderately certain can do), and 10 (certain can do). Total scores (ranging from 0-260) are calculated by summing the item scores and a higher score indicates higher coping self-efficacy.
Change in impact of traumatic life event | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  Impact Event Scale Revised (IES-R): The IES44 is a 15-item scale that assesses the impact of a traumatic life event, and has two subscales assessing the frequency of intrusive and avoidant cognitions associated with a specific stressor. It uses a 4-point scale, not at all to often to assess how often a respondent experienced specific symptoms during the past week. The IES was revised 45 to assess the three cluster symptoms of PTSD: intrusions, avoidance, and hyperarousal. Scores range from 0-88, with higher scores indicating more severe impact.
Change in post-traumatic stress disorder | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  Post-Traumatic Stress Disorder Checklist - Civilian Version (PCL-C): The PCL-C47 is a standardized 17-item self-report rating scale for PTSD. Respondents indicate how much they have been bothered by a symptom over the past month using a 5-point scale, with higher scores indicating more severe levels of PTSD, and it is a well-validated measure across different populations. Scores range from a minimum of 0, to a maximum of 80.
Change in post-traumatic growth | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  Post-Traumatic Growth Inventory (PTGI): The PTGI is a 21-item scale assessing positive outcomes reported by those who have experienced traumatic events.48 Items are scored on a 6-point scale and scores range from 0 to 105, with higher scores indicating greater levels of growth. It has good levels of internal consistency reliability (α=.90) and 2-month test-retest stability (r =.71).

OTHER OUTCOMES:
Socio-demographics | A. 24-48 hours before intervention (baseline)
  Data will be collected on the following: age, gender, marital status, highest level of education achieved, living situation (live alone, live with spouse, live with others), smoking status, alcohol/illicit drug use (yes, no; if yes, type and frequency of use), annual income after taxes, third-party insurance (yes, no), and employment status (employed, unemployed, retired, etc.), number/type of comorbid conditions, number/type of medications used by participant.
Injury Characteristics | A. 24-48 hours before intervention (baseline)
  The cause of injury will be obtained using the following categories: in a motor vehicle accident, hit by motor vehicle, fall, assault, stab, gunshot wound, recreational injury, and other. As well, whether the injury was unintentional, self-inflicted, assault, or cause unknown will be recorded.
Change in Injury Severity | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  Injury Severity Score (ISS): ISS49 assesses trauma severity, and correlates with mortality, morbidity and hospitalization time after trauma and is used to define the term 'major trauma'. ISS scores range from 0 to 75, and a major trauma is defined as an ISS being greater than 15.
Change in experiences in close relationships | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  Experiences in Close Relationships inventory-Short Form (ECR-S): The 12-item ECR-S evaluates the construct of adult attachment.50 Participants rate each of the 36 statements about connection using a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree). There is a minimum score of 7 and a maximum score of 42. Higher percentiles indicate more difficulty with attachment.
Change in Personality | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  Ten Item Personality Measure (TIPI): The TIPI assesses the Five-Factor Model of personality (agreeableness, neuroticism, conscientiousness, introversion, extraversion).52 It has adequate levels in terms of (a) convergence with widely used Big-Five measures in self, observer, and peer reports, (b) test-retest reliability, and (c) convergence between self and observer ratings.52 Each personality scale is measured on a scale of 1 (strongly disagree) to 7 ( strongly agree). Personality is an important determinant of outcome following injury as certain personality types may respond better to specific types of treatment,53 and has implications for the occurrence of PTSD.54
Reintegration | 3 months post-discharge
  Reintegration to Normal Living (RNL) Index: The RNL Index56 covers such areas as involvement in recreational and social activities, perceived ability to move within the community, and the degree of comfort people have with their relationships. It is a valid and reliable tool for assessing participation in various populations.56 Minimum score is 0 and maximum score is 100. Higher scores represent higher levels of participation.

CONTACTS AND LOCATIONS:
Overall Officials: Rosalie Steinberg, MSc, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nota SP, Bot AG, Ring D, Kloen P. Disability and depression after orthopaedic trauma. Injury. 2015 Feb;46(2):207-12. doi: 10.1016/j.injury.2014.06.012. Epub 2014 Jun 21. PMID 25015790
- [Background] Robinson LR. Trauma Rehabilitation. Lippincott Williams and Wilkins; 2006.
- [Background] Vranceanu AM, Bachoura A, Weening A, Vrahas M, Smith RM, Ring D. Psychological factors predict disability and pain intensity after skeletal trauma. J Bone Joint Surg Am. 2014 Feb 5;96(3):e20. doi: 10.2106/JBJS.L.00479. PMID 24500592
- [Background] Bandura A. Self-efficacy. The exercise of control. W.H. Freeman and Company; 1997.
- [Background] Connolly FR, Aitken LM, Tower M. An integrative review of self-efficacy and patient recovery post acute injury. J Adv Nurs. 2014 Apr;70(4):714-28. doi: 10.1111/jan.12237. Epub 2013 Sep 4. PMID 24001198
- [Background] Bosmans MW, van der Velden PG. Longitudinal interplay between posttraumatic stress symptoms and coping self-efficacy: A four-wave prospective study. Soc Sci Med. 2015 Jun;134:23-9. doi: 10.1016/j.socscimed.2015.04.007. Epub 2015 Apr 9. PMID 25875423
- [Background] Benight CC, Cieslak R, Molton IR, Johnson LE. Self-evaluative appraisals of coping capability and posttraumatic distress following motor vehicle accidents. J Consult Clin Psychol. 2008 Aug;76(4):677-85. doi: 10.1037/0022-006X.76.4.677. PMID 18665695
- [Background] Bei E, Kupeli N, Candy B. 47 The impact of supportive-expressive group therapy (SEGT) as an intervention on health-related outcomes and social support for people with advanced disease: a systematic review. BMJ Supportive & Palliative Care. 2018;8(3):377-378. doi:10.1136/bmjspcare-2018-mariecurie.47